CLINICAL TRIAL: NCT03817372
Title: Comparison of Anterior-Posterior Versus Anterior-Lateral Electrode Position in Cardioverting Atrial Fibrillation - A Randomized Clinical Trial
Brief Title: Electrode Positions in Cardioverting Atrial Fibrillation
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Viborg, Skive (Other); Randers Regional Hospital (Other); Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66051
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
Keywords: Cardioversion; Electrode position
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior-posterior electrode position (Active Comparator): The anterior electrode is placed in the left parasternal area (precordium). The posterior electrode is placed in the left lower-scapular region with the electrode edge left to the spinal column.
  Interventions: Device: Anterior-posterior electrode position
- Anterior-lateral electrode position (Active Comparator): The anterior electrode is placed in the right parasternal area below the clavicle. The lateral electrode is placed with the center of the electrode in the left mid-axillary line in level with the V6 electrocardiogram electrode.
  Interventions: Device: Anterior-lateral electrode position

INTERVENTIONS:
Device: Anterior-posterior electrode position — Escalating energy shocks (100 J, 150 J, 200 J, 360 J) using anterior-posterior electrode position
  Other Names: LIFEPAK 20, Physio-Control/Stryker
  Arms: Anterior-posterior electrode position
Device: Anterior-lateral electrode position — Escalating energy shocks (100 J, 150 J, 200 J, 360 J) using anterior-lateral electrode position
  Other Names: LIFEPAK 20, Physio-Control/Stryker
  Arms: Anterior-lateral electrode position

SUMMARY:
Atrial fibrillation is the most common heart rhythm disorder, and the incidence is rapidly increasing. Cardioversion using an electrical shock (DC-cardioversion) is an important treatment to reduce symptoms and improve patient's quality-of-life. The treatment is performed by applying gel electrodes to the chest. Cardioversion is not always successful, and it is unknown which electrode-position provides the optimal efficacy.

This study aims to compare two electrode positions, which are in clinical use: Anterior-posterior (left front and left back) versus anterior-lateral (right front and left side of the chest).

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation (documented on an ECG-12)
2. Able and willing to sign informed consent
3. Age ≥ 18 years
4. Anticoagulation according to guidelines (Patients with atrial fibrillation for >48 hours will be required to have a documented weekly international normalized ratio (INR) ≥2.0 (including within 48 hours of cardioversion) or treatment with non-vitamin K oral anticoagulant for three weeks or longer. Alternatively, a transoesophageal echocardiogram documenting the absence of intracardiac thrombi is accepted and cardioversion can be performed on treatment with low molecular weight heparin).

Exclusion Criteria:

1. Implanted pacemaker and/or cardioverter defibrillator (ICD)
2. Prior enrollment in the trial
3. Hemodynamically unstable atrial fibrillation
4. Untreated hyperthyroidism
5. Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Efficacy: First shock success | Immediately after first cardioversion attempt.
  The primary endpoint will be first shock efficacy, i.e. the proportion of patients in sinus rhythm for at least one minute immediately after an initial shock of 100 J.

SECONDARY OUTCOMES:
Efficacy: Successful cardioversion | One minute after cardioversion
  The secondary efficacy endpoint will be cardioversion success, i.e. the proportion of patients in sinus rhythm for at least one minute after end of protocol.
Safety: Number of participants with arrhythmic events during and after cardioversion | Within 2 hours after cardioversion (until discharge)
  Secondary safety endpoints will be arrhythmia during and after cardioversion (asystole, transient bradycardia, ventricular arrhythmia, atrioventricular block, recurrence of atrial fibrillation)
Safety: Number of participants with skin-discomfort, skin burns or itching | Two hours after cardioversion (at discharge)
  Patient-reported peri-procedural discomfort when asked at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Anders S Schmidt, MD, Principal Investigator — Randers Regional Hospital; Consultant cardiologist Andi E Albertsen, MD, PhD, Study Director — Viborg Regional Hospital; Professor Bo Løfgren, MD, PhD, FESC, FAHA, Study Chair — University of Aarhus
Locations (3):
- Denmark (3):
  - Horsens Regional Hospital, Horsens
  - Randers Regional Hospital, Randers
  - Viborg Regional Hospital, Viborg

REFERENCES:
- [Derived] Schmidt AS, Lauridsen KG, Moller DS, Christensen PD, Dodt KK, Rickers H, Lofgren B, Albertsen AE. Anterior-Lateral Versus Anterior-Posterior Electrode Position for Cardioverting Atrial Fibrillation. Circulation. 2021 Dec 21;144(25):1995-2003. doi: 10.1161/CIRCULATIONAHA.121.056301. Epub 2021 Nov 24. PMID 34814700